CLINICAL TRIAL: NCT04692948
Title: TAA6 Cell Injection In The Treatment of Patients With Relapsed / Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-TAA6-001
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: CAR; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAA6 cell injection (Experimental): Drug: TAA6 cell injection（Targeting CD276 autologous chimeric antigen receptor T cells）
  Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells.Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner, which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells.
  Interventions: Other: Chimeric antigen receptor T cells (car-t)

INTERVENTIONS:
Other: Chimeric antigen receptor T cells (car-t) — Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells. Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner, which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells.
  Other Names: TAA6 cell injection

SUMMARY:
This is a clinical study of TAA6 cell injection in the treatment of patients with relapsed / refractory Acute Myeloid Leukemia . The purpose is to evaluate the safety and effectiveness of CD276 targeted autologous chimeric antigen receptor T cells infusion in patients with relapsed / refractory CD276 positive Acute Myeloid Leukemia.（TAA6 cell injection is a T cell targeting CD276 chimeric antigen receptor）

DETAILED DESCRIPTION:
AML is a malignant disease of myeloid hematopoietic stem / progenitor cells and the most common hematological malignancy. It is characterized by abnormal proliferation of primitive and immature myeloid cells in bone marrow and peripheral blood. In recent years, due to the aging of the population, the incidence of AML and MDS has been on the rise. What is also troubling us is that the incidence of treatment-related MDS and AML in children and adolescents with Hodgkin's disease, sarcoma, breast and testicular tumors, lymphoma and other patients who survive after treatment is also gradually increasing. Occupational exposure such as ionizing radiation and benzene and petrochemical are also related to the incidence of AML.

Car t therapy is the most effective and widely used in the treatment of all. B7-H3, also known as cd276, was first discovered in 2001. It is mainly expressed on the cell surface, such as activated dendritic cells, monocytes, T cells, B cells and NK cells. Studies have shown that B7-H3 can stimulate the expansion and killing of T cells, and may selectively stimulate the signal receptor of T cells. It is a promising target for AML immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 (including the cut-off value), and the gender was not limited;
2. The expected survival time ≥ 12 weeks;
3. ECOG score 0-2;
4. After the standard treatment, the disease relapsed or progressed, and the researchers judged that there was no other positive effect Standard treatment plan;
5. The liver and kidney function and cardiopulmonary function meet the following requirements:

   1. Creatinine ≤ 1.5 ULN;;
   2. LVEF ≥ 45%;
   3. Blood oxygen saturation > 91%;
   4. Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN;
6. Able to understand the trial and have signed the informed consent.

Exclusion Criteria:

1. Patients with graft-versus-host disease (GVHD) or requiring immunosuppressive therapy;
2. In addition to cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical operation, and breast ductal carcinoma in situ after radical operation;
3. The patients with HBV (HCV) positive and HBV (HCV) positive in peripheral blood were detected for HBV (HCV) positive Syphilis was positive;
4. Severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥ III), severe arrhythmia;
5. Unstable systemic diseases judged by researchers: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
6. Within 7 days before screening, there were active or uncontrollable infections requiring systemic treatment (except mild urogenital infection and upper respiratory tract infection);
7. Pregnant or lactating women, female subjects planning pregnancy within 1 year after cell reinfusion or male subjects whose partners plan to conceive within 1 year after cell reinfusion;
8. Patients who had received car-t therapy or other gene modified cell therapy before screening;
9. Subjects who were receiving systemic steroid therapy within 7 days before screening or who were judged by the researcher to need long-term systemic steroid therapy during the treatment (except inhalation or local use);
10. Participated in other clinical studies within 3 months before screening;
11. There was evidence of central nervous system invasion during screening;
12. According to the judgment of the researchers, it does not conform to the condition of cell preparation;
13. Other researchers think that it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
ORR 3 ORR 3 | three months after CAR-T cells infusion
  3-month objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, Principal Investigator — No.1, Swan Lake Road, new administrative and Cultural District, Hefei City, Anhui Province
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China